CLINICAL TRIAL: NCT02610179
Title: Strawberry Candy Twists as an Alternative Screen for Gestational Diabetes: A Prospective Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Kjersti Aagaard, Associate Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: H-35564
Record Dates: First submitted 2015-11-13; First posted 2015-11-20 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Glucola GCT (Active Comparator): A prospective cohort of 617 women who will undergo screening for gestational diabetes with the standard glucola GCT between 24 and 28 weeks gestational age.
  Interventions: Dietary Supplement: Standard Glucola GCT
- Twizzlers challenge (Experimental): At a later date, the same prospective cohort of 617 women Participants will receive their Twizzlers challenge between 24 and 28 weeks gestational age.
  Interventions: Dietary Supplement: Twizzlers challenge

INTERVENTIONS:
Dietary Supplement: Standard Glucola GCT — Participants will be screened with the standard method of consumption of the glucola beverage followed by a 1 hour venous blood draw.
  Arms: Standard Glucola GCT
Dietary Supplement: Twizzlers challenge — Participants will consume the Twizzlers equivalent (10 strawberry flavored Twizzlers) and have their venous blood glucose checked in 1 hour.
  Arms: Twizzlers challenge

SUMMARY:
The goal of this prospective study is to determine whether there is superiority of 10 Twizzlers to the 50 gram glucola beverage for screening for GDM in a population based study.

DETAILED DESCRIPTION:
The aim now is to perform a large, prospective trial to test Twizzlers® as a cost effective glucola alternative in a gravid population to determine its sensitivity, specificity, PPV (positive predictive value) and NPV (negative predictive value) alongside ROC (receiver operating curve) from a population-based cohort.

Participants will be enrolled among the pregnant patients in the Harris Health System Obstetrics Clinics who are either due for the standard glucola GCT (glucose challenge test) or who have had their glucola screening but have not had the 3 hour GTT (glucose tolerance test). These women will be offered the opportunity to consume the Twizzler equivalent of the 50 gm glucola beverage (10 strawberry flavored Twizzlers) and to have their venous blood glucose checked 1 hour post consumption. This will all be done while the patient is in clinic and will not necessitate any extra clinic visits on their behalf. They will then go on to be scheduled for their confirmatory 3 hour glucose tolerance tests if indicated by any abnormality in either their glucola GCT or their Twizzlers challenge. The efficacy of Twizzlers will then be compared to the 50 gm glucola beverage as a screen for gestational diabetes. Specifically, the sensitivity, specificity, PPV, NPV, NNT (number needed to treat), ROC, and referral rates for each mode of screening will be calculated.

For the Twizzler portion of the study, the subjects will consume 10 strawberry Twizzlers within 5 minutes. One hour after consumption begins each participant will have a blood draw to check a serum glucose level. Within the same day, the samples will be delivered to Dr. Morey Haymond's lab for analysis.

Serum glucose and insulin levels will be tested on each sample. The amount of each blood sample will be approximately 10 ml of blood (2 teaspoons). Sample collection (blood draws; venipuncture) will allow for testing the serum glucose levels of subjects after consumption of Twizzlers. These values will be used for analysis to determine if Twizzlers are truly equivalent to the Glucola beverage. Ultimately, the patient's will only undergo 1 extra venipuncture than what they would have had as part of their routine prenatal care if both screening tests are normal. There is a possibility of undergoing a 3 hour GTT that would not have otherwise been performed if the subjects Twizzlers screen is elevated but glucola was normal.

Participants will receive a phone call to report any abnormal values on their GCT as per standard clinical operating measures, and will have their GTT scheduled with the nursing staff. Based on prior studies, a notable rate of false-positives is not anticipated with the Twizzler GCT. In the rare occasion that such occurs (i.e., screen positive by Twizzler but not by glucola beverage) they will be informed of the need for a 3 hour GTT. This will be covered by the study costs, and their insurance will not be charged.

Pregnancy outcomes data for subjects will be collected, including gestational age at delivery, mode of delivery and any complications, maternal weight gain, and infant birthweight. This will all be acquired as data abstraction from the EMR and maintained in a secure coded database.

Otherwise, there will be no further contact or requirements of the subject.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* 24 to 28 weeks gestation
* Singleton or twin or triplet gestation
* Willing to participate in the study

Exclusion Criteria:

* Known Type II DM
* Known Type I DM
* On oral or injectable corticosteroids
* 50 gram glucola beverage GCT of greater than or equal to 190 mg/dl

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 617 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The serum glucose levels will be measured in response to oral glucose challenge and compared between Twizzlers and glucola beverage. | 24 to 28 weeks gestation
  Each participant will have a blood draw to check the serum glucose level.

SECONDARY OUTCOMES:
Cost-effectiveness | 24 to 28 weeks gestation
  The cost-effectiveness of Twizzlers over the glucola beverage will be measured in a small gravid cohort by taking into account the cost per unit of Twizzlers versus glucola.

CONTACTS AND LOCATIONS:
Overall Officials: Kjersti Aagaard, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Ben Taub General Hospital, Houston, Texas, United States